CLINICAL TRIAL: NCT06966739
Title: Multispectral Optoacustic Imaging in Patients With Myositis
Acronym: MYOMSOT
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: MYOMSOT
Record Dates: First submitted 2025-03-12; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Myositis
Keywords: msot; medical treatment; myositis; functional parameters
MeSH Terms: conditions — Myositis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myositis: Patients with myositis should be included as well as healthy age and sex matched individuals als control group.
  Interventions: Other: MSOT of musculature

INTERVENTIONS:
Other: MSOT of musculature — All measurements using multispectral optoacustic tomography (MSOT) are performed on the paraspinal muscles as well as the trapezius, rectus abdominus and the proximal and distal limb muscles in a right vs. left comparison (leg proximal: quadriceps and ischiocrural muscle, leg distal triceps surae muscle, tibialis anterior muscle; arm proximal: M. biceps, distal: forearm flexors).

SUMMARY:
Myositis syndromes are a relatively rare group of diseases in which acquired inflammation of the muscles occurs. According to clinical, histological and immunopathological criteria, autoimmune (dermatomyositis, polymyositis, immune-mediated necrotizing myopathy, anti-synthetase syndrome, inclusion body myositis), pathogen-related and so-called special forms (e.g. checkpoint-inhibitor-related) of myositis can be distinguished.

A typical symptom of the disease is progressive muscle weakness. In addition, especially a possible extramuscular organ manifestation can lead to increased morbidity.

The initiation of appropriate drug therapy and regular follow-ups to measure the success of the therapy are of crucial importance. Magnetic Resonance Imaging (MRI) and sonography are imaging methods that have proven effective for this purpose to date.

The former can be used to detect changes such as fatty remodeling, edema or inflammatory changes using T1- and T2-weighted images and Short-Tau-Inversion-Recovery (STIR). However, the duration of the examination, the lack of space and the high costs are certainly a limitation of the examination. Furthermore, patients with corresponding contraindications, such as a pacemaker.

Sonography of the musculature is therefore also important. In particular, changes in the muscle parenchyma in the sense of increasing echogenicity can be detected in this context. Moreover, regional atrophy can also be detected in this modality. However, myosonography is more of a screening procedure for neuromuscular diseases than it is suitable for monitoring progression and therapy.

Another option is the method of multispectral optoacoustic imaging (MSOT), in which ultrasound is combined with optical imaging using laser beams.

Depending on the wavelength, different chromophores such as hemoglobin or melanin (wavelength in the visible range of light) or lipids and proteins (wavelength in the near-infrared range, long-wave light) can be imaged.

Optoacoustic imaging thus provides information about morphological as well as molecular and functional conditions.

The advantages of this imaging have already been established in the context of various neuromuscular diseases:

For example, a significant increase in collagen concentration was shown in patients with Duchenne muscular dystrophy compared to a healthy control group as a possible marker of fibrosis. A significant correlate was also found in the clinical neurological examination. Particularly striking here was an indirect correlation between the 6-minute walk test and the collagen concentration.

The aforementioned imaging can also offer advantages for patients with neuromuscular diseases, particularly with regard to therapy monitoring.

Objective and quantitative measurement of disease progression is essential here. Optoacoustic imaging allows functional and molecular parameters in particular to be differentiated. This enables early and objective quantitative measurement of possible tissue loss, which can ultimately influence further therapy.

The aim of the present study is to carry out functional and molecular imaging using optoacoustic imaging to evaluate possible functional and molecular parameters, which may prove to be suitable markers for monitoring progression.

The aim of the study is to investigate whether the examination technique could be suitable for monitoring the progression of myositis.

All patients with a neuromuscular disease of the NMZ will be included in this trial.

ELIGIBILITY:
Inclusion Criteria:

* patients with myositis undergoing treatment at the integrated muscle center (imz) of the University Hospital of Gießen

Exclusion Criteria:

* contraindications against an optoacoustic examination
* pregnancy
* ingestion of photosensitizers within the last 72 hours
* current phototherapy
* known photosensitive disorder

Min Age: 18 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consits of patients with myositis and an age and gender matched control group.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Parchenchmymal changes in the muscles in the context of myositis | From enrollment to the end of examinations six months
  The primary endpoint of the study is the concentration of hemoglobin as correlate for an ongoing inflammation in the muscle compared to a healthy control group. The following hypothesis applies: The concentration of hemoglobin is increased in patients with myositis compared to a healthy control group.

SECONDARY OUTCOMES:
Concentration of collagen and lipids in the musculature compared to a healthy control group | From enrollment to the end of examinations six months
  Myositis is known to lead to remodelling processes in the muscles, in the sense of connective tissue or fatty remodelling. Therefore, the secondary outcome parameter is the concentration of collagen in the musculature of patients with myositis compared to a healthy control group. A further secondary outcome measure is the concentration of lipids in the muscles of patients with myositis as a correlate for fatty remodelling.
  It is hypothesised that the concentration of lipids and collagen is increased in patients with myositis compared to a healthy control group.

CONTACTS AND LOCATIONS:
Overall Officials: Heidrun Krämer-Best, Prof. Dr., Study Chair — Uniklinik Giessen
Locations (1):
- Justus-Liebig-Universität Gießen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided